CLINICAL TRIAL: NCT04855604
Title: A Cross-sectional Study on the Status Quo of Diagnosis and Treatment of Pediatric Outpatients With Respiratory Diseases in China
Brief Title: The Status Quo of Diagnosis and Treatment of Pediatric Outpatients With Respiratory Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Baoping XU, Chief of Respiratory Department Affiliation: Beijing Children's Hospital, Beijing Children's Hospital
Other Study IDs: BCH Lung 015
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Respiratory Diseases
Keywords: respiratory diseases; treatment; medication; children
MeSH Terms: conditions — Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study is expected to conducted by inquiring about the history, diagnosis results and medication details of respiratory diseases of the outpatient pediatric patients with respiratory diseases in the pediatric departments at specialist children's hospital at the second class and above, general hospitals and maternal and child healthcare hospitals. About 10,000 electronic questionnaires are expected to be collected in total, with about 100 participating hospitals and 100 electronic questionnaires from each participating hospital.Diagnosis and treatment information of pediatric patients are expected to be collected in the third week in April, July and October 2021 and in January 2022.

DETAILED DESCRIPTION:
Respiratory diseases are easy-to-transmit among and are common in children, especially acute respiratory infections in children which contribute to more than 60% of pediatric outpatient cases. In pediatric internal medicine outpatient cases, trachitis/bronchitis, acute upper respiratory tract infection, pneumonia, acute tonsillitis and asthma are the most common diseases torturing pediatric patients.

Children are prone to recurrent respiratory infections which may impose heavy burdens on their families. Ten million children under 5 years old are killed by recurrent respiratory infections every year. In China, daily outpatient visits of children with recurrent upper respiratory tract infections account for 10%-20% of the total daily outpatient visits for respiratory diseases. The outpatient medication for pediatric patients is found of non-compliance issues. According to the data in 2014, more than 33.8% of pediatric patients of all ages were given off-label medication, and more than 30% were given off-label medication in treatment.

The trial will be completed in 1 years with 10,000 participants taken from hospitals in partnership with clinical research collaboration of National Clinical Research Center for Respiratory Diseases, China, and analyze the status quo of diagnosis results and medication details of respiratory diseases of the outpatient pediatric patients with respiratory diseases in China.

ELIGIBILITY:
Inclusion Criteria:

* All children participating in this clinical study must meet all of the following criteria.

  1. age: 0-14 years old, male and female;
  2. accord with diagnostic criteria of respiratory diseases
  3. Agreed to informed consent

Exclusion Criteria:

* All children with any of the following conditions must be excluded from this study:

  1. children who visit hospital duo to discharge of hospital
  2. Children who visit hospital beyond 2 times in 7 days.

Ages: 1 Day to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children aged between 0-14 years, and diagnosed with respiratory disease can be enrolled in our study with their (or their parents') agreements.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
General information of pediatric patients | 1 year
  General information of pediatric patients

SECONDARY OUTCOMES:
History of respiratory diseases and medication of pediatric patients in the past year | 1 year
Diagnosis and medication information of pediatric patients in the Study | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Baoping Xu, Beijing, Beijing Municipality, China